CLINICAL TRIAL: NCT01924403
Title: Assessment of Wound Closure Techniques in Primary Total Knee Arthroplasty Using SPY Intra-operative Angiography
Brief Title: Perfusion Assessment of Wound Closure Techniques in Primary Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Robert T. Trousdale, Professor of Orthopedic Surgery, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-005083
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Total Knee Arthroplasty
Keywords: TKA; Wound Closure; Wound Perfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Staple Closure (Experimental): Staple closure will be one technique employed to close the wound in primary total knee arthroplasty.
  Interventions: Procedure: Staple Closure
- Running Subcuticular Closure (Experimental): Running subcuticular closure will be one technique employed to close the wound in primary total knee arthroplasty.
  Interventions: Procedure: Running Subcuticular Closure
- Vertical Mattress Closure (Experimental): Vertical mattress closure will be one technique employed to close the wound in primary total knee arthroplasty.
  Interventions: Procedure: Vertical Mattress Closure

INTERVENTIONS:
Procedure: Staple Closure
  Arms: Staple Closure
Procedure: Vertical Mattress Closure
  Arms: Vertical Mattress Closure
Procedure: Running Subcuticular Closure
  Arms: Running Subcuticular Closure

SUMMARY:
This study will assess which of the three most common methods of wound closure in primary total knee arthroplasty (staples, interrupted vertical mattress, or running subcuticular suture) provide the best wound vascular perfusion. This can be achieve by using SPY intra-operative vascular angiography, which is commonly used in clinical practice to assess perfusion of wound closure at the clinic. By understanding the differences in perfusion afforded by different closure techniques, surgeons will then be able to select the technique that optimizes this parameter so as to avoid complications such as tissue necrosis, wound dehiscence, or infection.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Primary diagnosis of osteoarthritis
* Surgical indication for index total knee arthroplasty

Exclusion Criteria:

* Previous surgery about the knee
* Systemic corticosteroid use
* Active infection of any kind or chronic infection with HIV, Hepatitis C, or Syphilis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Perfusion of Wound Closure | Surgical Point of Care

CONTACTS AND LOCATIONS:
Overall Officials: Robert Trousdale, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Wyles CC, Jacobson SR, Houdek MT, Larson DR, Taunton MJ, Sim FH, Sierra RJ, Trousdale RT. The Chitranjan Ranawat Award: Running Subcuticular Closure Enables the Most Robust Perfusion After TKA: A Randomized Clinical Trial. Clin Orthop Relat Res. 2016 Jan;474(1):47-56. doi: 10.1007/s11999-015-4209-x. PMID 25733009